CLINICAL TRIAL: NCT06018402
Title: The Effect of Erector Spinae Plane Block in Combination With Physical Therapy on Pain, Disability, and Quality of Life in Patients With Degenerative Scoliosis: Prospective, Randomized, Clinical Study
Brief Title: The Effect of Physical Therapy Program and Erector Spina Plane Block in Patients With Degenerative Lumbar Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozge Illeez, MD, Principal Investigator, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ozgeilleez1
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: Degenerative lumbar scoliosis; Physical treatment; Erector spinae plane block; Low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Prospective, Randomised, Clinical Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy (Active Comparator): The physical therapy program is planned as a total of 15 sessions in the lumbar region, each session consisting of TENS (50-100 Hz stimulation frequency, 200 µs pulse duration, intensity is increased as much as the patient could tolerate, 20 minutes in total), hotpack (to be placed on the painful area, 20 minutes), US (1 mHz frequency, 10 minutes, 1.5 watt/cm2 intensity)
  Interventions: Other: physical therapy
- physical therapy + espb (Active Comparator): same physical therapy program, in addition Ultrasound-guided lumbar ESPB is performed using an in-line cephalic approach, and after contacting the corner of the L3 transverse process, a small dose of saline is injected into the fascial space between the L3 transverse process and the erector spinae muscles to "lift off" the fascia. After verification, a mixture of 20 mL of 1% lidocaine and 3 mg betamethasone is administered for unilateral injection. The procedure is performed bilaterally.
  Interventions: Other: physical therapy + espb

INTERVENTIONS:
Other: physical therapy — The physical therapy program is planned as a total of 15 sessions in the lumbar region, each session consisting of TENS (50-100 Hz stimulation frequency, 200 µs pulse duration, intensity is increased as much as the patient could tolerate, 20 minutes in total), hotpack (to be placed on the painful area, 20 minutes), US (1 mHz frequency, 10 minutes, 1.5 watt/cm2 intensity).
  Arms: physical therapy
Other: physical therapy + espb — the same physical therapy program, in addition Ultrasound-guided lumbar ESPB is performed using an in-line cephalic approach, and after contacting the corner of the L3 transverse process, a small dose of saline is injected into the fascial space between the L3 transverse process and the erector spinae muscles to "lift off" the fascia. After verification, a mixture of 20 mL of 1% lidocaine and 3 mg betamethasone is administered for unilateral injection. The procedure is performed bilaterally.
  Arms: physical therapy + espb

SUMMARY:
Degenerative (de novo) scoliosis is the result of a long and multifactorial process that occurs through degenerative change in the aging population without a pre-existing spinal deformity. Pain is the most important symptom and the major difference from adolescent idiopathic scoliosis. Treatment is often complex and patient-specific. The first aim of our study is to evaluate the effectiveness of physical therapy on pain, disability and quality of life in patients with degenerative lumbar scoliosis and the second aim is to investigate whether erector spina plan block (ESPB) combined with physical therapy has an effect on the results.

DETAILED DESCRIPTION:
Patients over 60 years of age, with low back or low back-leg pain for at least 3 months, who had received pharmacologic treatment but did not respond, and diagnosed with degenerative lumbar scoliosis are included in the study. Patients are randomized into to groups according to the interventions as: physical therapy group (G-1) and physical therapy and ESPB injection group (G-2). The physical therapy program is planned as a total of 15 sessions in the lumbar region, each session consisting of TENS (50-100 Hz stimulation frequency, 200 µs pulse duration, intensity is increased as much as the patient could tolerate, 20 minutes in total), hotpack (to be placed on the painful area, 20 minutes), US (1 mHz frequency, 10 minutes, 1.5 watt/cm2 intensity). Ultrasound-guided lumbar ESPB is performed using an in-line cephalic approach, and after contacting the corner of the L3 transverse process, a small dose of saline is injected into the fascial space between the L3 transverse process and the erector spinae muscles to "lift off" the fascia. After verification, a mixture of 20 mL of 1% lidocaine and 3 mg betamethasone are administered for unilateral injection. The procedure is performed bilaterallyThe primary endpoint of the study is pain intensity assasment by using a numerical rating scale (NRS), and secondary endpoints are functional status, quality of life and disability status assasment by using SRS-22 and Oswestry disability index. Patients are evaluated before and 1 week, 1 month and 3 months after treatment. In the 2nd group, pain intensity at 1 hour after injection is additionally evaluated with a NRS. As a result of the power analysis, the minimum sample size was planned as a total of 16 patients with 8 patients in each group with a 15% dropout rate. Shapiro Wilk test is applied to examine the normality of the data distribution. The difference between groups is evaluated by Mann Whitney U according to normal distribution and by ANOVA for time-dependent within-group change.

ELIGIBILITY:
Inclusion Criteria:

* Being 60 years or older
* Having a scoliosis of 10 degrees or more in the lumbar region according to the measurement made with the cobb method
* Having pain in the axial waist or radiating from the waist to the leg
* Pain that persists for at least 3 months
* NRS > 4

Exclusion Criteria:

* Systemic or local infection at the injection site
* Past or current history of malignant disease
* Presence of neurological or orthopedic disease
* Presence of uncontrolled hypertension, diabetes mellitus
* Presence of severe heart failure
* Presence of bleeding diathesis
* Anticoagulant use
* Lidocaine allergy
* Psychiatric disorder or mental problem
* inflammatory spine pain
* Severe osteoporosis / previous vertebral fracture
* Body mass index >35
* Having had previous surgery on the lumbar region
* Injection was applied to the waist region within 6 months or physical have been treated

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
NRS (Numeric Rating Scale) | Day 0
  Pain Intensity Assessment ( 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS (Numeric Rating Scale) | 1 hour after injection
  Pain Intensity Assessment ( 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS (Numeric Rating Scale) | 1 week after physical treatment
  Pain Intensity Assessment ( 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS (Numeric Rating Scale) | 1 month after physical treatment
  Pain Intensity Assessment ( 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS (Numeric Rating Scale) | 3 month after physical treatment
  Pain Intensity Assessment ( 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
SRS-22 | Day 0
  22 questions make up the SRS-22, which covers five domains: function/activity, pain, self-perceived image, mental health, and satisfaction with therapy. Scores range from 1 (worst) to 5 (best) for each item.
SRS-22 | 1 week after physical treatment
  22 questions make up the SRS-22, which covers five domains: function/activity, pain, self-perceived image, mental health, and satisfaction with therapy. Scores range from 1 (worst) to 5 (best) for each item.
SRS-22 | 1 month after physical treatment
  22 questions make up the SRS-22, which covers five domains: function/activity, pain, self-perceived image, mental health, and satisfaction with therapy. Scores range from 1 (worst) to 5 (best) for each item.
SRS-22 | 3 month after physical treatment
  22 questions make up the SRS-22, which covers five domains: function/activity, pain, self-perceived image, mental health, and satisfaction with therapy. Scores range from 1 (worst) to 5 (best) for each item.
Oswestry Disability Index | Day 0
  Each item has six statements and is scored between 0 and 5. The overall score is then calculated as a percentage, with 0% denoting no disability and 100% denoting the highest level of disability, with 0 denoting the least disability and 5 denoting the worst.
Oswestry Disability Index | 1 week after physical treatment
  Each item has six statements and is scored between 0 and 5. The overall score is then calculated as a percentage, with 0% denoting no disability and 100% denoting the highest level of disability, with 0 denoting the least disability and 5 denoting the worst.
Oswestry Disability Index | 1 month after physical treatment
  Each item has six statements and is scored between 0 and 5. The overall score is then calculated as a percentage, with 0% denoting no disability and 100% denoting the highest level of disability, with 0 denoting the least disability and 5 denoting the worst.
Oswestry Disability Index | 3 month after physical treatment
  Each item has six statements and is scored between 0 and 5. The overall score is then calculated as a percentage, with 0% denoting no disability and 100% denoting the highest level of disability, with 0 denoting the least disability and 5 denoting the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Gulsum Illeez, Study Director — Fatih Sultan Mehmet Taining and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Farih Sultan Mehmet Training and Research Hospital, Istanbul
  - Fatih Sultan Mehmet Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham RB, Sugrue PA, Koski TR. Adult Degenerative Scoliosis. Clin Spine Surg. 2016 Apr;29(3):95-107. doi: 10.1097/BSD.0000000000000367. PMID 26945131
- [Background] Ploumis A, Transfledt EE, Denis F. Degenerative lumbar scoliosis associated with spinal stenosis. Spine J. 2007 Jul-Aug;7(4):428-36. doi: 10.1016/j.spinee.2006.07.015. Epub 2007 Feb 28. PMID 17630141
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Ahiskalioglu A, Alici HA, Ciftci B, Celik M, Karaca O. Continuous ultrasound guided erector spinae plane block for the management of chronic pain. Anaesth Crit Care Pain Med. 2019 Aug;38(4):395-396. doi: 10.1016/j.accpm.2017.11.014. Epub 2017 Dec 15. No abstract available. PMID 29253539
- [Background] Akyuz ME, Firidin MN. Bilateral ultrasound-guided erector spinae plane block for postoperative persistent low back pain in lumbar disc surgery. Eur Spine J. 2022 Jul;31(7):1873-1878. doi: 10.1007/s00586-022-07212-z. Epub 2022 Apr 14. PMID 35420380
- [Background] Durmus IE, Surucu S, Muz A, Takmaz SA. The effectiveness of erector spinae plane block in patients with chronic low back pain. Eur Rev Med Pharmacol Sci. 2023 Jan;27(1):138-143. doi: 10.26355/eurrev_202301_30864. PMID 36647861